CLINICAL TRIAL: NCT06096116
Title: Phase 3, Double-blind, Placebo-controlled, Multicentre Study on the Efficacy and Safety of Human Plasma Derived Antithrombin (Atenativ) in Heparin-Resistant Patients Scheduled to Undergo Cardiac Surgery Necessitating Cardiopulmonary Bypass
Brief Title: Phase 3 Study on the Efficacy and Safety of Human Plasma Derived Antithrombin (Atenativ) in Heparin-Resistant Patients Scheduled to Undergo Cardiac Surgery Necessitating Cardiopulmonary Bypass
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATN-108
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acquired Antithrombin Deficiency
Keywords: heparin resistance; antithrombin deficiency; cardiopulmonary bypass; cardiac surgery
MeSH Terms: conditions — Antithrombin III Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) The patients, care provider administering IMP, and outcomes assessors will be blinded from treatment allocations. Delegated study personnel preparing the IMP will be unblinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-dose Atenativ (Experimental): Patients will receive a single bolus of 30 international units (IU)/kg body weight (BW) Atenativ.
  Interventions: Drug: Human plasma derived antithrombin
- High-dose Atenativ (Experimental): Patients will receive a single bolus of 60 international units (IU)/kg body weight (BW) Atenativ.
  Interventions: Drug: Human plasma derived antithrombin
- Placebo (Placebo Comparator): Patients will receive a saline bolus dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human plasma derived antithrombin — A solvent/detergent and heat-treated antithrombin concentrate derived from human plasma
  Arms: High-dose Atenativ; Low-dose Atenativ
Drug: Placebo — Half of the patients in the placebo group will be randomised to receive a volume of placebo corresponding to the low dose of Atenativ and the other half to receive a volume of placebo corresponding to a high dose of Atenativ
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of two different doses of Atenativ, versus placebo, in restoring and maintaining heparin responsiveness in adult patients undergoing cardiac surgery necessitating cardiopulmonary bypass (CPB)

ELIGIBILITY:
Inclusion Criteria:

1. Planned cardiac surgery with CPB
2. Heparin-resistant patients (pre-CPB Hemochron ACT less than 480 s in the measurement taken between 2-5 minutes following intravenous administration of 500 U/kg UFH)
3. Patients between 18 and 85 years of age, inclusive
4. Freely given written or electronic informed consent
5. In female patients of childbearing potential, a pre-existing negative pregnancy test within 14 days prior to surgery

Exclusion Criteria:

1. Receiving, or have received within the timeframes specified, one or more of the following medications prior to the start of surgery:

   1. vitamin K antagonists (within 3 days)
   2. direct oral anticoagulants (within 2 days)
   3. thienopyridines (ticlopidine within 14 days, prasugrel within 7 days, or clopidogrel within 5 days), unless platelet function is satisfactory according to local standard of care assessment
   4. ticagrelor (within 5 days), unless platelet function is satisfactory according to local standard of care assessment
   5. glycoprotein IIb/IIIa antagonist (within 24 hours)
2. Pre-existing coagulopathy, a history of bleeding problems, or a laboratory-diagnosed bleeding disorder (e.g., von Willebrand disease, platelet disorder)
3. Renal insufficiency, defined as serum creatinine level >2.0 mg/dL
4. Thrombocytosis, defined as platelet count >400,000 per μL
5. Known hypersensitivity or allergic reaction to antithrombin or any of the excipients in Atenativ, i.e., human albumin, sodium chloride, acetyl tryptophan, caprylic acid
6. History of anaphylactic reaction(s) to blood or blood components
7. Refusal to receive transfusion of blood or blood-derived products
8. Current participation in another interventional clinical trial or previous participation in the current trial
9. Treatment with any IMP within 30 days prior to screening visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Restoring heparin responsiveness | During surgery (from the time of the first surgical incision to the time at which the final suture or staple is placed)
  The percentage of patients in each group in whom no further therapy containing antithrombin (i.e. frozen plasma or other antithrombin concentrates) is needed for restoring pre-CPB heparin responsiveness after administration of Atenativ or placebo, and for maintaining it during CPB

SECONDARY OUTCOMES:
Amounts of further therapy for restoring heparin responsiveness | During surgery (from the time of the first surgical incision to the time at which the final suture or staple is placed)
  The comparison between the amounts of further therapy containing antithrombin (i.e., FP or antithrombin concentrates) needed for restoring pre-CPB heparin responsiveness, after administration of Atenativ or placebo, and for maintaining it during CPB
Change in activated clotting time (ACT) values | Within 5 minutes following intravenous administration of 500 U/kg unfractionated heparin (UFH) and between 2-10 minutes after IMP infusion
  The comparison between the change in ACT values following infusion of each of the Atenativ doses and placebo
Change in antithrombin plasma levels | Within 10 minutes before IMP infusion and between 2 and 10 minutes after IMP infusion, within 10 minutes after the end of CPB, at the end of surgery, and at 24 hours after the start of IMP infusion
  The comparison between the change in antithrombin plasma levels following infusion of each of the Atenativ doses and placebo
Change in heparin usage | From end of IMP infusion to the end of surgery
  The comparison between heparin usage following the infusion of each of the Atenativ doses and infusion of placebo
FP unit use | From the start of IMP infusion until 24 hours following IMP infusion, and until discharge or 7 days after surgery, whichever comes first
  The comparison between the number of units of FP transfused for reasons other than restoring or maintaining heparin responsiveness, both intraoperatively (from the start of Atenativ or placebo infusion until the start of CPB, during CPB, and from the end of CPB until the end of surgery) and postoperatively (from the end of surgery until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first), as well as cumulatively
Amounts of further antithrombin concentrate for maintaining heparin responsiveness | From placement of the final suture or staple until 24 hours following IMP infusion, to discharge or 7 days after surgery, whichever comes first
  The comparison between postoperative use of antithrombin concentrates for reasons other than restoring heparin responsiveness (from the end of surgery until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first)
Transfusion of allogenic blood products | From the start of IMP infusion until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first
  The comparison between transfusion of other allogeneic blood products (e.g., red blood cells [RBCs], platelets, cryoprecipitate, whole blood, albumin, other transfusion), both intraoperatively (from the start of Atenativ or placebo infusion until the start of CPB, during CPB, and from the end of CPB until the end of surgery) and postoperatively (from the end of surgery until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first), as well as cumulatively
Administration of coagulation factor concentrates | From the start of IMP infusion until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first
  The comparison between administration of coagulation factor concentrates (fibrinogen concentrate, factor XIII concentrate, recombinant activated factor VII, other therapy)", both intraoperatively (from the start of Atenativ or placebo infusion until the start of CPB, during CPB, and from the end of CPB until the end of surgery) and postoperatively (from the end of surgery until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first), as well as cumulatively
Administration of other haemostatic-relevant therapies | From the start of IMP infusion until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first
  The comparison between administration of other haemostatic-relevant therapies (i.e., tranexamic acid, aminocaproic acid, protamine, other therapies), both intraoperatively (from the start of Atenativ or placebo infusion until the start of CPB, during CPB, and from the end of CPB until the end of surgery) and postoperatively (from the end of surgery until 24 hours after the start of Atenativ or placebo infusion and until discharge or 7 days after surgery, whichever comes first), as well as cumulatively
Postoperative chest tube drainage | From the start of IMP infusion to 24 hours after infusion and until discharge or 7 days after surgery, whichever comes first
  The comparison between postoperative chest tube drainage volume at 24 hours after the start of Atenativ or placebo infusion, and the comparison between total chest tube drainage volume until discharge or 7 days after surgery, whichever comes first
Need for reoperation due to bleeding | 24 hours after the start of IMP infusion
  Comparison of the need for reoperation for bleeding, including description of the cause of bleeding (surgical vs. non-surgical)
Cell saver volume | During surgery (from the time of the first surgical incision to the time at which the final suture or staple is placed)
  The comparison between cell saver volume until the end of surgery
Adverse events | From the start of IMP infusion until hospital discharge or 7 days after IMP administration, whichever comes first
  Incidence of adverse events, including all related and non-related, non-serious adverse events
Serious adverse events | From the start of IMP infusion until 28 days after IMP administration
  Incidence of serious adverse events
Survival status | At hospital discharge or 7 days after IMP administration (whichever comes first) and at 28 days (+ 4 days) after IMP administration
  Number of patients surviving in all three cohorts
Red Blood Cell count | Within 10 minutes before IMP infusion, between 2-10 minutes after IMP infusion, within 10 minutes after the end of CPB, at the end of surgery, and at 24 hours after infusion
  Standard haematological parameter
White Blood Cell count | Within 10 minutes before IMP infusion, between 2-10 minutes after IMP infusion, within 10 minutes after the end of CPB, at the end of surgery, and at 24 hours after infusion
  Standard haematological parameter
Haemoglobin levels | Within 10 minutes before IMP infusion, between 2-10 minutes after IMP infusion, within 10 minutes after the end of CPB, at the end of surgery, and at 24 hours after infusion
  Standard haematological parameter
Haematocrit | Within 10 minutes before IMP infusion, between 2-10 minutes after IMP infusion, within 10 minutes after weaning from CPB, at the end of surgery, and at 24 hours after infusion
  Standard haematological parameter
Platelet count | Within 10 minutes before IMP infusion, between 2-10 minutes after IMP infusion, within 10 minutes after weaning from CPB, at the end of surgery, and at 24 hours after infusion
  Standard haematological parameter

CONTACTS AND LOCATIONS:
Locations (24):
- United States (8):
  - Stanford University School of Medicine, Stanford, California
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - OU Health University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Austria (2):
  - University Hospital Innsbruck, Innsbruck
  - Vienna General Hospital AKH, Medical University of Vienna, Vienna
- Canada (4):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- Czechia (2):
  - Center of Cardiovascular and Transplant Surgery, Brno
  - Institute for Clinical and Experimental Medicine, Prague
- France (2):
  - CHU de Reims, Hôpital Robert Debré, Reims
  - CHU de Rennes, Rennes
- Hospital of Lithuanian university of Health sciences Kauno Klinikos, Kaunas, Lithuania
- Institute for Cardiovascular Diseases C.C. Iliescu, Bucharest, Romania
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- United Kingdom (3):
  - Royal Papworth Hospital, Cambridge
  - University Hospital Coventry and Warwickshire, Coventry
  - The James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: No